CLINICAL TRIAL: NCT02352805
Title: A Comparative Clinical Study to Understand the Coagulopathy and Systemic Inflammation Associated With the Use of Extracorporeal Circulation in Intensive Care Patients
Brief Title: Coagulopathy and SIRS During ECC in Intensive Care
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: COSIMA
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Disorder of Circulatory System
Keywords: Extracorporeal circulation, ventricular assist device

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human whole blood and blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- (1) veno-venous ECMO: ECMO - Patients being connected to veno-venous extracorporeal membrane oxygenation (ECMO)
  Interventions: Device: ECLS/ECC
- (2) veno-arterial ECLS: ECLS - Patients being connected to veno-arterial extracorporeal life support (ECLS)
  Interventions: Device: ECLS/ECC
- (3) LVAD (Heart Mate II): LVAD - Patients being connected to a left ventricular assist device (LVAD) (Heart Mate II)
  Interventions: Device: ECLS/ECC
- (4) LVAD (Heart Ware): LVAD - Patients being connected to a left ventricular assist device (LVAD) (Heart Ware)
  Interventions: Device: ECLS/ECC
- (5) LVAD (Impella): LVAD - Patients being connected to a left ventricular assist device (LVAD) (Impella)
  Interventions: Device: ECLS/ECC
- (6) Dialysis system: Patients being connected to a dialysis system
  Interventions: Device: ECLS/ECC
- (7) LVAD (Heart Mate III): LVAD - Patients being connected to a left ventricular assist device (LVAD) (Heart Mate III)
  Interventions: Device: ECLS/ECC
- (8) HLM: HLM = Heart Lung Machine - patients undergoing coronary artery bypass grafting surgery and / or aortic valve replacement with cardiopulmonary bypass
  Interventions: Device: ECLS/ECC

INTERVENTIONS:
Device: ECLS/ECC — Extracorporeal circulation and mechanical circulatory support for heart or lung or renal failure during intensive care therapy or cardiac surgery

SUMMARY:
This observational clinical study investigates cellular and plasmatic activation markers as well as proteins involved in coagulation and inflammation in patients being connected to different extracorporeal circulation (ECC) and circulatory support devices under intensive care conditions.

DETAILED DESCRIPTION:
The complex interplay between the various factors contributing to the ECC-related coagulopathy and inflammation in intensive care settings is only poorly understood so far. Furthermore, it is unclear, how coagulopathy and inflammation shall be monitored and which anticoagulants may be employed to decrease complications associated with specific ECC systems. Therefore, the use of laboratory analyses, anticoagulation and anti-platelet therapy varies between different ECC systems and intensive care units.

A better understanding of the mechanisms of the activation and interaction of platelets and leukocytes, plasmatic coagulation, complement, cytokines and endothelium will highlight starting-points to increase the safety and efficacy of ECC in intensive care medicine. The investigation of these phenomena in different ECC systems under clinical conditions is therefore the goal of this study.

In order to achieve the study goal, we will investigate cellular and plasmatic activation markers as well as proteins involved in coagulation and inflammation in patients being connected to different ECC systems under intensive care conditions.

ELIGIBILITY:
Inclusion Criteria:

Need for therapy with extracorporeal circulation / circulatory support due to cardiac failure, or lung failure, or renal failure, or a combination of these diseases

Exclusion Criteria:

1. History of previously diagnosed hereditary coagulation and/or platelet disorders
2. Refusal to receive blood transfusion
3. Participation in other clinical research studies involving evaluation of other investigational drugs or devices within 30 days of randomization
4. Diagnosis of hepatitis B, hepatitis C, and HIV
5. Age > 85 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients undergoing implantation of extracorporeal circulation or mechanical circulatory support systems (ECLS / ECMO / LVAD / dialysis) due to cardiac failure, or lung failure, or renal failure, or a combination of these diseases.
  * Patients undergoing cardiac surgery with extracorporeal circulation (ECC).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of the platelet activation marker "beta-thromboglobulin" | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Helene Häberle, MD, Principal Investigator — University of Tübingen, Dept. of Anesthesiology and Intensive Care Medicine, Germany
Locations (1):
- Dept. of Anesthesiology and Intensive Care Medicine, University Hospital Tübingen, Tübingen, Germany